CLINICAL TRIAL: NCT06171282
Title: A Clinical Safety and Efficacy Study on Oncolytic Virus Injection (R130) for the Treatment of Advanced Bone and Soft Tissue Tumors
Brief Title: A Clinical Study on Oncolytic Virus Injection (R130) for the Treatment of Advanced Bone and Soft Tissue Tumors
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Shanghai Yunying Medical Technology (Industry)
Collaborators: Shanghai General Hospital, Shanghai Jiao Tong University School of Medicine (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SHYY-R130-BSTT
Record Dates: First submitted 2023-12-06; First posted 2023-12-14 (Actual); Last update posted 2023-12-14 (Actual); Status verified 2023-12

CONDITIONS: Osteosarcoma; Sarcoma; Soft Tissue Sarcoma; Bone Tumor
Keywords: Oncolytic virus; Herpes simplex virus type 1; Immunotherapy
MeSH Terms: conditions — Osteosarcoma; Sarcoma; Bone Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental: R130 Treatment Group (Experimental): Every 7-14 days,1-2 ml R130 （concentration of 1x10^8 plaque-forming Units/mL,PFU/mL）will be injected intratumoral in patients with relapsed/refractory bone and soft tissue tumors.
  Interventions: Drug: Recombinant oncolytic herpes simplex virus type Ⅰ (R130)

INTERVENTIONS:
Drug: Recombinant oncolytic herpes simplex virus type Ⅰ (R130) — R130, a modified herpes simplex virus-Ⅰ (HSV-1) containing the gene coding for anti-CD3 scFv/CD86/PD1/HSV2-US11
  Other Names: Oncolytic virus Injection

SUMMARY:
9 participants are expected to be enrolled for this open，Single-armed clinical trial to evaluate the safety and efficacy of the recombinant herpes simplex virus Ⅰ, R130 in patients with advanced bone and soft tissue tumors.

ELIGIBILITY:
Inclusion Criteria:

1. Age 16 to 75 years, diagnosed with soft tissue sarcoma or bone neoplasms clearly by histology and/or cytology.
2. Failure of standard treatment or patient unwillingness to receive other antitumor therapy.
3. No absolute or relative centasis contraindiction.
4. Subjects with ECoG score of 0-2.
5. Expected survival of 3 months or more.
6. Have at least one measurable lesion (according to RECIST 1.1 criteria) that is amenable to intratumoral drug delivery.
7. Subjects must have appropriate organ function, and laboratory tests during the screening period must meet the following requirements: a) absolute neutrophil count (ANC) ≥ 1.5 × 109/L, platelets (PLT) ≥ 80 × 109/L, and hemoglobin (Hb) ≥ 85 g/L; b) serum creatinine (Cr) and blood urea nitrogen (BUN) within 1.5 times the upper limit of normal values; c) serum total bilirubin (TBIL) ≤ 2 times the upper limit of normal values; d) glutamic aminotransferase (ALT) and glutamic oxalacetic aminotransferase (AST) ≤ 2.5 times the upper limit of normal values; subjects with liver metastases do not exceed 5 times the upper limit of normal values; e) activated partial thromboplastin time (APTT), prothrombin time (PT) within 1.5 times the upper limit of normal values.
8. Any treatment for malignancy, including radiotherapy, chemotherapy and biological agents, must be discontinued 28 days prior to R130 treatment.
9. Eligible patients of childbearing potential must agree to use a reliable method of contraception (hormonal or barrier method or abstinence) with their partner for the duration of the trial and for at least 180 days after the last dose; female patients of childbearing potential must have a negative urine pregnancy test within 7 days prior to enrollment.
10. Subjects voluntarily sign an informed consent form and are in good compliance.

Exclusion Criteria:

1. Have had any serious adverse reactions associated with immunotherapy and have not recovered to CTCAE 5.0 grade rating 0 or 1 level of toxicity after previous antineoplastic therapy.
2. Subjects with any severe and/or uncontrolled disease, including: a) poorly controlled hypertension (systolic blood pressure ≥ 150 mmHg or diastolic blood pressure ≥ 100 mmHg); b) suffering from class I or higher myocardial ischemia or myocardial infarction, arrhythmia (QTc ≥ 470 ms and ≥ grade 2 congestive heart failure (New York Heart Association (NYHA) classification); c) active or uncontrolled severe infection (≥ CTCAE grade 2 infection); d) Patients with previous organ transplantation, bone marrow transplantation (hematopoietic stem cell transplantation) and severe immune deficiency; e) Urine routine suggesting urine protein ≥++ and confirmed 24-hour urine protein quantification > 1.0 g.
3. Patients with past history of type I diabetes mellitus or HIV.
4. Severe abnormalities in thyroid and cortisol testing; active, known or suspected autoimmune disease requiring systemic therapy.
5. Patients with active tuberculosis and a strong positive OT test.
6. Patients with active bleeding or severe coagulation dysfunction.
7. Have had antitumor therapy, including endocrine, chemotherapy, radiotherapy, targeted therapy, immunotherapy and antitumor herbal therapy, 4 weeks prior to the first dose.
8. Current active hepatitis B, active hepatitis C, immunodeficiency virus or other active infection of clinical significance.
9. Patients who have undergone surgery of grade 3 or higher or whose surgical wounds have not healed within 4 weeks prior to enrollment.
10. Pregnant, lactating and planning to have children within six months.
11. Subjects who, in the judgment of the investigator, are unsuitable for participation in this trial for any reason.

Ages: 16 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 9 (Estimated)
Dates: Start 2023-07-12 (Actual); Primary Completion 2025-07-12 (Estimated); Study Completion 2026-07-12 (Estimated)

PRIMARY OUTCOMES:
Subject incidence of adverse events | Up to 6 months
  To characterize the safety profile of R130 injection in patients with relapsed/refractory bone and soft tissue tumors as measured by the incidence of Grade ≥ 3 Common Terminology Criteria for Adverse Events, version 5.0 (CTCAE v5.0)
Subject incidence of laboratory abnormalities | Up to 1 month
  Detection of liver and renal function, electrocardiogram, routine blood examination etc
Systemic Immune Response | Up to 6 months
  Detection of increased systemic immune Response markers in sera (IL2,IL4,IL6,IL8,IL10,TNFa，IFNγ, etc.) and peripheral blood mononuclear cells by multi-Color fluorescence-activated cell sorting (FACS)

SECONDARY OUTCOMES:
Disease Assessment for Disease Control Rate | Every 10 weeks for 12 months
  Evaluate the efficacy endpoints of DCR by the investigator with RECIST v1.1 and iRECIST
Disease Assessment for Duration of Response | Every 10 weeks for 12 months
  Evaluate the efficacy endpoints of DOR by the investigator with RECIST v1.1 and iRECIST
Quality of Life Assessment | Every 6 weeks for 12 months
  Evaluate with EORTC QLQ-C30

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai General Hospital, Shanghai, China

IPD SHARING:
Plan to Share IPD: Undecided